CLINICAL TRIAL: NCT03930641
Title: An Open-Label, Single-Arm, Multicenter, Phase IIIb Study in Patients With Neovascular Age-Related Macular Degeneration to Evaluate the Safety of Brolucizumab 6 mg in Prefilled Syringe
Brief Title: Study of the Safety of Brolucizumab 6 mg in Prefilled Syringe in Patients With Neovascular Age Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258A2308
Record Dates: First submitted 2019-04-26; First posted 2019-04-29 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-07

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: brolucizumab 6 mg prefilled syringe PFS; open label study; neovascular age related macular degeneration intravitreal injection IVT; observation
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: study with a single arm: brolucizumab 6 mg PFS
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RTH258 (Experimental): brolucizumab 6 mg in a prefilled syringe
  Interventions: Drug: RTH258

INTERVENTIONS:
Drug: RTH258 — 6 mg in prefilled syringe
  Other Names: brolucizumab

SUMMARY:
This was a multicenter, open label study that is designed to evaluate the safety of brolucizumab 6 mg in a prefilled syringe in subjects with neovascular age related macular degeneration and to support collection of observations of the prefilled syringe use for intravitreal injection.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety of brolucizumab 6 mg delivered in a pre-filled syringe (PFS) in subjects with neovascular age-related macular degeneration (nAMD) with the primary endpoint being the incidence of ocular and non-ocular adverse events (AEs). There were no other objectives for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Study eye is diagnosed with neovascular age related macular degeneration and would need an intravitreal injection.
3. Subjects >= 50 years of age.

Exclusion Criteria:

1. Active infection or inflammation in the eyes.
2. Uncontrolled glaucoma.
3. History of a medical, ocular or non-ocular conditions, resulting in that the study medication cannot be safely administered.
4. Treatment with anti-VEGF intravitreal injection in the study eye within one month prior to enrollment.
5. The use of intraocular corticosteroids in the study eye within the last three months prior to enrollment.
6. Recent intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation.
7. Uncontrolled hypertension.

Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Novartis Investigative Site, Altamonte Springs, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of the patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five subjects were enrolled and 34 received one IVT injection of brolucizumab 6 mg PFS. One subject withdrew consent before receiving treatment.
Period: Overall Study
Arm/Group | RTH258
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RTH258
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.9 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Brolucizumab 6 mg Delivered in Prefilled Syringe in Patients With Neovascular Age Related Macular Degeneration
Description: The safety is defined as the incidence of ocular and non-ocular adverse events
Time Frame: Up to Day 31
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | RTH258
Number analyzed (Participants) | 34
Participants
  Adverse Events | 0
  Deaths | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 post treatment, up to maximum duration of approximately two months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. Normal reporting of treatment emergent AEs which are not SAEs are normally reported with an incidence greater than or equal to 5%.
Arm/Group | RTH258
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03930641/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03930641/SAP_001.pdf